CLINICAL TRIAL: NCT04314479
Title: Improving Adherence to American Cancer Society (ACS) Guidelines on Nutrition and Physical Activity Through Integrated Symptom Management in Latinas With Cancer and Their Informal Caregivers
Brief Title: Improving Adherence to ACS Guidelines on Nutrition and Physical Activity in Latinas With Cancer and Their Informal Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1801209654
Record Dates: First submitted 2020-03-16; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Cancer
Keywords: Cancer; Cancer symptoms; Cancer survivors; Latina; Nutrition; Healthy lifestyle
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptom Assessment and Health Coaching (Experimental): The intervention condition will involve weekly symptom assessment and health coaching to manage symptoms and to meet the ACS cancer prevention guidelines provided over the telephone by trained health coaches. Participants will be completing the same forms/assessments throughout the study. The content will be built around the Symptom Management Toolkit. The coaching will be dictated by the symptoms the survivor or the support person is experiencing the week of the intervention call. All calls begin with the symptom assessments, only the intervention arm includes intervention coaching that focuses on physical activity, stress management, or eating a healthy diet to improve adherence to the ACS guidelines for cancer prevention. We anticipate coaching sessions will last approximately 20 - 45 minutes
  Interventions: Behavioral: Symptom Assessment and Health Coaching
- Symptom Assessment Only (Other): For participants randomized to the control condition weekly symptom assessment telephone calls will be completed by staff at the University of Arizona Cancer Center Behavioral Measurements Interventions Shared Resource (BMISR). At week 13 an exit interview will be completed by the study coordinator to record participants feedback regarding study intervention, length, coaches, etc… In addition, staff from BMISR will call to repeat all baseline measures with the exception of the demographic questionnaires. Symptom assessment calls will take approximately 15 minutes.
  Interventions: Behavioral: Symptom Assessment and Health Coaching

INTERVENTIONS:
Behavioral: Symptom Assessment and Health Coaching — The intervention condition will involve weekly symptom assessment and health coaching to manage symptoms and to meet the ACS cancer prevention guidelines provided over the telephone by trained health coaches. Participants will be completing the same forms/assessments throughout the study. The content will be built around the Symptom Management Toolkit. The coaching will be dictated by the symptoms the survivor or the support person is experiencing the week of the intervention call. All calls begin with the symptom assessments, only the intervention arm includes intervention coaching that focuses on physical activity, stress management, or eating a healthy diet to improve adherence to the ACS guidelines for cancer prevention. We anticipate coaching sessions will last approximately 20 - 45 minutes.

SUMMARY:
This research study is testing the feasibility and acceptability of a 12-week intervention that integrates telephone coaching and printed materials about the ACS guidelines and healthy lifestyle behaviors in order to manage symptoms after treatment for cancer. We will recruit 57 dyads (the survivor plus one identified informal caregiver) from the community.

DETAILED DESCRIPTION:
This research study is testing the feasibility and acceptability of a 12-week intervention that integrates telephone coaching and printed materials about the ACS guidelines and healthy lifestyle behaviors in order to manage symptoms after treatment for cancer. The study population is 36 Latinas who have recently completed treatment for solid tumor cancers and their informal caregiver (36 dyads). Research suggests that family members can be facilitators to behavior change more specifically, Latinos rely on family support more than non-Hispanic Whites.

Fewer than 20% of Latina cancer survivors meet the American Cancer Society's (ACS) Guidelines on Nutrition and Physical Activity. Healthier lifestyle behaviors (such as diet and physical activity) would result in an immediate benefit of reduced symptoms and long-term benefit of improved health while lowering cancer risk. This pilot study tests an intervention that will help in lessening survivors' symptoms to improve adherence to the ACS guidelines for cancer prevention ultimately improving overall health. A telephone-based intervention does not require any in-person meetings (outside of initial recruitment) and lessens participant burden.

The Specific Aims of this project are to evaluate this intervention among 36 survivors who have recently completed treatment for solid tumor cancers and their informal caregivers to 1) Determine the feasibility and acceptability of the intervention 2) Establish the preliminary efficacy for improvement in diet, physical activity, and quality of life for the dyads, and symptom burden for survivors through surveys given at baseline and study completion as well as a weekly symptom distress survey.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Female
* at least 18 years of age
* diagnosis of cancer
* speak and understand English or Spanish
* are finishing (or have finished) curative intent cancer treatment and do not have any subsequent cancer treatments planned, except for hormonal therapy or trastuzumab for breast cancer.
* Patients must also have at least 1 of the 5 most common cancer-related symptoms (pain, sleep disturbance, anxiety, depression and/or fatigue) with a severity score of 4 or higher (2 or higher for depression) on a 0-10 rating scale which is based on the National Comprehensive Cancer Network guidelines for symptom monitoring.

Caregivers

* must be 18 years or older
* able to speak and understand English or Spanish
* not currently treated for cancer preserving the distinction between survivor and caregiver.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must be female; caregiver may be male or female
Enrollment: 144 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2019-06-16 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility | 12 weeks
  Feasibility assessed by consent rate of 50% and 2) completion rate of intervention of 80% Acceptability assessed by open-ended questions as part of exit interview/satisfaction survey at end of study (80% benchmark for dyads considering intervention helpful).
Determine acceptability | 12 weeks
  Acceptability assessed by completion rate of intervention of 80%. Acceptability assessed by open-ended questions as part of exit interview/satisfaction survey at end of study (80% benchmark for dyads considering intervention helpful).
Establish preliminary efficacy in diet adherence. | 12 weeks
  Preliminary efficacy for improvement assessed utilizing NCI Dietary Screener Questionnaire for diet.
Establish preliminary efficacy in physical activity adherence. | 12 weeks
  Preliminary efficacy for improvement assessed utilizing Women's Health Initiative (WHI) Physical Activity Questionnaire for physical activity.
Establish preliminary efficacy via symptom improvement. | 12 weeks
  Preliminary efficacy for improvement assessed utilizing General Symptom Distress Scale for symptoms/QoL and Patient Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy Short Form for self-efficacy for symptom management.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy E. Crane, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No